CLINICAL TRIAL: NCT04650464
Title: Cardiopulmonary Fitness in Children With Asthma Versus Healthy Children : VO2 Asthma
Brief Title: Cardiopulmonary Fitness in Children With Asthma Versus Healthy Children
Acronym: VO2asthma
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0022
Record Dates: First submitted 2020-10-07; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-10

CONDITIONS: Asthmatic
Keywords: Asthmatic children; VO2 max; Physical fitness; Peadiarics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma is the most common chronic disease in children worldwide. Asthma is characterised by a chronic inflammatory disorder of the airways,episodes of wheezing, breathlessness, chest tightness and coughing. There is a large variability of asthma prevalence between countries from 11 to 15% for children in developed countries.

Asthma may limit the patient's ability to be physically active and can lead to a sedentary lifestyle and affect patients' quality of life. Indeed, long-term goal of asthma management as any chronic disease is to control symptoms in order to ensure a normal quality of life to children with asthma In 1980, the World Health Organization stated that functional capacity explorations best reflect the impact of a chronic disease on the quality of life. Indeed, cardiopulmonary exercise test (CPET) has become the "gold standard" in functional evaluation of cardiorespiratory diseases in adults gradually extended to children. Physical fitness is evaluated by maximal oxygen uptake "VO2 max" during a CPET. CPET also allows to determine possible limiting factors (cardiac limitation, ventilatory limitation, muscular deconditioning) responsible for a lower VO2max.

There is actually contradictory evidence regarding the aerobic fitness levels of asthmatic children and it remains unclear whether significant differences exist between asthmatic children and their non-asthmatic counterparts. Few studies suggest ventilatory exercise limitations linked to the severity of bronchial obstruction whether others put in light the impact of muscular deconditioning in the asthmatic population.

In this context, the investigators aimed to compare the cardiopulmonary fitness of children with asthma with that of age-adjusted and gender-adjusted controls. The investigators also intended to identify clinical characteristics associated with VO2max in this population.

DETAILED DESCRIPTION:
This retrospective study was carried out from November 2010 to September 2015 for control children (already published PMID: 29170358) : and January 2015 to December 2019 for asthmatic children.

CPET were realised in 2 paediatric CPET laboratories (centre 1: Montpellier University Hospital, France; centre 2: Paediatric Cardiology and Rehabilitation Centre, Institut-Saint-Pierre, Palavas-Les-Flots, France).

Children aged 5 to 18 years old were recruited in one of the 2 CPET laboratories.

Two groups were identified: children with asthma and the control children.

1. The asthma group consisted of children followed for asthma by any pediatrician or pulmonologist and referred to one of the 2 CPET laboratories. The following clinical data were collected : gender, weight, height, treatments to deduce treatment level (GINA step), associated pathologies, activity level, symptoms during exercice
2. The control group consisted of children referred for a non-severe functional symptom linked to exercise (murmur, palpitation, or dyspnoea) or for a medical sports certificate. These children were classified in the control group only after a completely normal check-up, including physical examination, electrocardiogram, echocardiography, and spirometry. Children with any chronic disease, medical condition (cardiac, neurologic, respiratory, muscular, or renal), or medical treatment and those requiring any further specialized medical consultation were not eligible. The clinical data collected concerned gender, weight, height.

CPET procedures in both centres were harmonized before the study started. Spirometry was systematically performed before the exercise test with a flow volume curve and measurement of forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and the FEV1/FVC ratio (FEV1/FVC), with normalization to GLI 2012 Z scores. The same investigator coordinator manually calculated the VO2max and the ventilatory anaerobic threshold (VAT) using Beaver's method. VO2max and VAT values were normalized in a percentage of the predicted VO2max using normal values from Wasserman and Cooper. The investigators considered VO2max below 80% of predicted value as pathologic value and a VAT value below 55 % of predicted VO2max was in favor of muscular deconditioning.

All informations from CPET were recorded : heart rate (HR), blood pressure (BP), estimated VO2/HR, VAT, breathing reserves (BR), respiratory rate (RR), VE/VCO2 slope, Tidal Volume (VT)

ELIGIBILITY:
Inclusion criteria:

* Children aged 5 to 18 years old recruited in one of the 2 CPET laboratories after a regular paediatric cardiology outpatient visit.
* The asthma group consisted of children followed for asthma by any pediatrician or pulmonologist and referred to one of the 2 CPET laboratories.
* The control group consisted of children referred for a non-severe functional symptom linked to exercise (murmur, palpitation, or dyspnoea) or for a medical sports certificate.

Exclusion criteria:

* patients <5 years or 1,2m, patients >18 ans
* absolute contraindications : fever, uncontrolled asthma, respiratory failure, acute myocarditis or pericarditis, uncontrolled arrhythmias causing symptoms or haemodynamic compromise, uncontrolled heart failure, acute pulmonary embolus or pulmonary infarction, and children with mental impairment leading to inability to cooperate
* parents refuse the use of medical data
* for the control group : children with any chronic disease, medical condition (cardiac, neurologic, respiratory, muscular, or renal), medical treatment, requiring any further specialized medical consultation or with any finding at clinical and paraclinical examination (electrocardiogram, echocardiography)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 5 to 18 years old recruited in one of the 2 CPET laboratories after a regular paediatric cardiology outpatient visit.
  Cases : children with asthma Control : healthy children from a cohort already published (PMID: 29170358)
Sampling Method: Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison cardiopulmonary fitness in children with asthma versus healthy children | 1 day
  Comparison VO2max in children with asthma versus healthy children.

SECONDARY OUTCOMES:
Comparison of others CPET in children | 1 day
  Comparison of others CPET in children with asthma versus healthy children
Variation of VO2max in asthmatic children | 1 day
  Clinical and functional factors associated with lower VO2max in asthmatic children

CONTACTS AND LOCATIONS:
Overall Officials: Johan Moreau, MD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Moreau J, Socchi F, Renoux MC, Requirand A, Abassi H, Guillaumont S, Matecki S, Huguet H, Avesani M, Picot MC, Amedro P. Cardiopulmonary fitness in children with asthma versus healthy children. Arch Dis Child. 2023 Mar;108(3):204-210. doi: 10.1136/archdischild-2021-323733. Epub 2022 Nov 29. PMID 36446481